CLINICAL TRIAL: NCT00828464
Title: An Open Label Study to Evaluate Safety, Efficacy and Tolerability of Clobetasol Propionate for the Condition of Chronic Hand Dermatitis
Brief Title: Study to Evaluate Safety, Efficacy and Tolerability of Clobetasol Propionate for Chronic Hand Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stiefel, a GSK Company (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Organization: GlaxoSmithKline (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: U0280-401
Record Dates: First submitted 2009-01-22; First posted 2009-01-26 (Estimated); Results first posted 2010-09-28 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-09

CONDITIONS: Hand Dermatosis
Keywords: Dermatosis, Dermatitis, Dry skin, Irritated skin
MeSH Terms: conditions — Hand Dermatoses; Skin Diseases; Dermatitis | interventions — Clobetasol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- clobetasol propionate foam (Experimental): All subjects receive clobetasol propionate
  Interventions: Drug: clobetasol propionate

INTERVENTIONS:
Drug: clobetasol propionate — Clobetasol propionate. The study product will be applied topically twice a day (morning and evening) for 14 days of treatment.

SUMMARY:
The purpose of the study is to assess the safety, efficacy and tolerability of Clobetasol propionate foam in subjects with chronic dermatitis.

DETAILED DESCRIPTION:
The study is being conducted in order to obtain safety, efficacy and tolerability data for Clobetasol propionate foam in the treatment of chronic dermatitis. The subjects must have mild to moderate disease based on the Investigator's assessment at baseline.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 18 years of age or older, with diagnosis of chronic dermatitis, able to complete the study and comply with study instructions.
* Female subjects of childbearing potential must have a negative pregnancy test. Sexually active women of childbearing potential participating in the study must have been using a medically acceptable form of contraception

Exclusion Criteria:

* Use of systemic corticosteroid and/or other prohibited medications within 4 weeks of the baseline visit.
* Use of topical corticosteroid therapy and/or other prohibited topical medications within 2 weeks prior to the baseline visit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Physicians Skin Care, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Kircik LH, Tropmann C. Treatment of mild-to-moderate chronic hand dermatitis with clobetasol propionate 0.05% EF foam: results from an open-label study. J Drugs Dermatol. 2011 Dec;10(12):1398-402. PMID 22134563

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * Recruitment period: First Subject Enrolled October 2008, Last Subject Enrolled January 2009.
  * Type of location: Dermatology Research Center
Pre-assignment Details: 1. Washout from use of systemic corticosteroid and/or other prohibited medications if used within 4 weeks of the baseline visit.
  2. Washout from use of topical corticosteroid therapy and/or other prohibited topical medications if used within 2 weeks prior to the baseline visit
Groups:
- Clobetasol Propionate Foam: All subjects applied clobetasol propionate 0.05% foam twice a day (morning and evening) to the hands.
Period: Overall Study
Arm/Group | Clobetasol Propionate Foam
Started | 30
Completed | 29
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 30
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 47.5 (14.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Region of Enrollment [Number; unit: participants]
  United States | 30
ISGA-Chronic Hand Dermatitis [Number; unit: Participants] — Investigators Static Global Assessment (ISGA)- Chronic Hand Dermatitis Score=2 mild Score=3 moderate These are the only scores that are permitted for entry on this study.
  Participants
    Mild | 16
    Moderate | 14
Time since Diagnosis of Chronic Hand Dermatitis (years) [Mean (Standard Deviation); unit: Years] — Time since Diagnosis of Chronic Hand Dermatitis, Allergic, Irritant or Contact Dermatitis (years)
  Years | 18.92 (15)
Total Hand Eczema Severity Index (HESI) [Mean (Standard Deviation); unit: Units on a scale] — Total Hand Eczema Severity Index (total HESI) Score 0 to 360 where 0 is the best and 360 is the worst score.
  Units on a scale | 32.1 (17.0)

OUTCOME MEASURES:

1. Secondary Outcome: Proportion of Subjects Who Achieve at Least a 1-grade Improvement Based on the ISGA at Day 8.
Description: Please note that the proportion of participants is being reported as a percentage of participants.
  Investigator's Static Global Assessment Score (ISGA) At least 1-grade improvement (%) at Day 8
  ISGA grades:
  Score = 0 (Clear) Score = 1 (Almost Clear) Score = 2 (Mild) Score = 3 (Moderate) Score = 4 (Severe)
Time Frame: Baseline, Day 8
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 76.7

2. Primary Outcome: Proportion of Subjects With at Least 1-grade Improvement From Baseline to Day 15 in Investigator's Static Global Assessment Score (ISGA) Score
Description: Proportion of Subjects with at least a 1-Grade Improvement from Baseline to Day 15 In Investigator's Static Global Assessment Score (ISGA) - Chronic Hand Dermatitis Please note that the proportion of participants is being reported as a percentage of participants.
  ISGA grades:
  Score = 0 (Clear) Score = 1 (Almost Clear) Score = 2 (Mild) Score = 3 (Moderate) Score = 4 (Severe)
Time Frame: Baseline, Day 15
Population: Intent-to-treat (ITT).
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 96.7

3. Secondary Outcome: Change in Subject's Visual Analogue Assessment Scale
Description: Mean change in subject's visual analogue assessment scale from baseline to day 8. At each visit, the subject is requested to rate the changes in their skin on the hands on a 1 to 10 scale with 0 being poor and 10 being excellent.
Time Frame: Baseline, Day 8
Population: ITT. Twenty-nine of the 30 subjects enrolled on this study had results for this endpoint on day 8. Thirty of the 30 subjects enrolled had results for this same assessment at the day 15 visit.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 29
Units on a scale | 1.46 (2.25)

4. Secondary Outcome: Proportion of Subjects at Day 15 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Finger Tips
Description: Proportion of subjects at day 15 with at least 1-Grade improvement in the Hand Eczema Severity Index Score (HESI) for all symptoms present at baseline - Finger Tips. The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 15
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 73.3

5. Secondary Outcome: Proportion of Subjects at Day 8 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Finger Tips
Description: Proportion of Subjects at day 8 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Finger Tips
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 8
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 43.3

6. Secondary Outcome: Proportion of Subjects at Day 15 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline - Fingers
Description: Proportion of Subjects at day 15 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Fingers.
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 15
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 70

7. Secondary Outcome: Proportion of Subjects With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Fingers
Description: Proportion of Subjects at day 8 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline - Fingers
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 8
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 50

8. Secondary Outcome: Proportion of Subjects at Day 8 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Palm of Hands
Description: Proportion of Subjects at Day 8 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline - Palm of Hands.
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 8
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 56.7

9. Secondary Outcome: Proportion of Subjects at Day 15 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Palm of Hands
Description: Proportion of Subjects at Day 15 with at least a 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Palm of Hands The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 15
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 73.3

10. Secondary Outcome: Proportion of Subjects at Day 8 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Back of Hands
Description: Proportion of Subjects at Day 8 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Back of Hands.
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 8
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 33.3

11. Secondary Outcome: Proportion of Subjects at Day 15 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Back of Hands
Description: Proportion of Subjects at Day 15 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Back of Hands.
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 15
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 66.7

12. Secondary Outcome: Proportion of Subjects at Day 8 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Wrists
Description: Proportion of Subjects at Day 8 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Wrists.
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 8
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 40

13. Secondary Outcome: Proportion of Subjects at Day 15 With at Least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI) for All Symptoms Present at Baseline Wrists
Description: Proportion of Subjects at Day 15 with at least 1-Grade Improvement In the Hand Eczema Severity Index Score (HESI)for All Symptoms Present at Baseline Wrists.
  The proportion of participants is being reported as a percentage of participants.
  Each hand was divided into five areas [fingertips, fingers (except the tips), palms, back of hands and wrists]. For each of these areas the intensity of the 6 following clinical signs: erythema, induration, papulation, vesicles, fissuring, scaling and oedema was graded as follows: 0, no skin changes; 1, mild disease; 2, moderate and 3, severe.
Time Frame: Baseline, Day 15
Population: ITT
Measure: Number; unit: Percentage of Participants
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Percentage of Participants | 40

14. Secondary Outcome: Change in Subject's Visual Analogue Assessment Scale From Baseline to Day 15
Description: Mean change in subject's visual analogue assessment scale from baseline to day 15. At each visit, the subject is requested to rate the changes in their skin on the hands on a 1 to 10 scale with 0 being poor and 10 being excellent.
Time Frame: Baseline, Day 15
Population: ITT
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Clobetasol Propionate Foam
Number analyzed (Participants) | 30
Units on a scale | 3.40 (2.50)

ADVERSE EVENTS:
Time Frame: 15 days
Arm/Group | Clobetasol Propionate Foam
Serious Adverse Events (participants affected / at risk) | 1/30
Other Adverse Events (participants affected / at risk) | 4/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol Propionate Foam (N=30)
Skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clobetasol Propionate Foam (N=30)
Application site burning (General disorders) | 2 (2)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Open label study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days